CLINICAL TRIAL: NCT04376151
Title: Acceptance and Commitment Therapy Guided Self-help for Adults With a Diagnosis of Autistic Spectrum Disorder Experiencing Psychological Distress
Brief Title: Guided ACT and for Adults With ASD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lincoln (Other)
Collaborators: Nottinghamshire Healthcare NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 245597
Record Dates: First submitted 2020-02-24; First posted 2020-05-06 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Autism Spectrum Disorder (ASD)
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: The intervention is a guided self-help Acceptance and Commitment Therapy (ACT) bibliotherapy, written by Steven Hayes called 'Get Out of your Mind and Into Your Life'. This book has been split into eight sections, participants will be asked to read one section each week. Each week each participant will speak with the researcher to ask any questions and review the weeks material via a guided telephone call. All telephone calls will follow a pre-determined list of questions to increase standardisation and recorded for fidelity checks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants will work through an Acceptance and Commitment Therapy informed self-help bibliotherapy over a period of eight weeks. The bibliotherapy is called 'Get Out of Your Life and Into your Mind' written by Steve. C. Hayes.
  Interventions: Other: Acceptance and Commiment Therapy (ACT) bibliotherapy 'Get Out of Your Mind and Into Your Life'

INTERVENTIONS:
Other: Acceptance and Commiment Therapy (ACT) bibliotherapy 'Get Out of Your Mind and Into Your Life' — The intervention has been described in the arm/group descriptions.

SUMMARY:
This study aims to investigate the efficacy of guided self-help Acceptance Commitment Therapy (ACT) for adults who have a diagnosis for Autistic Spectrum Disorder (ASD) and are experiencing psychological distress (stress, anxiety or depression).

This is a repeated measures design, using a single case experimental design (SCED) over a period of fourteen weeks. Each participant (n=8) with be asked to complete weekly measures and shortened measures every three days, while they read an ACT guided self-help bibliotherapy. For more information about the measures, please see outcome measure section. The ACT guided bibliotherapy will be administered to each participant on a weekly basis, over eight weeks.

Participants will be asked to complete outcome measures at two week and at four weeks post intervention.

DETAILED DESCRIPTION:
INTRODUCTION High levels of psychiatric co-morbidity have been found with adults who receive a diagnosis of Autistic Spectrum Disorder (ASD); including stress, anxiety, depression and OCD.

Acceptance and Commitment Therapy (ACT) is a psychotherapeutic approach and is referred to as a "third wave" CBT. There have been over one hundred randomized control trials (RCTs) supporting the efficacy of ACT for different types of distress and severity. Researchers conducted an ACT based group, for students with ASD; the results indicated that levels of stress, hyperactivity and emotional distress were reduced in the treatment group, compared to classes as unusual. Results were maintained or improved at a two month follow up. However, little is still known about the efficacy of ACT for adults with ASD who experience.

This research will indicate if guided ACT self-help facilitates increases psychological flexibility for adults with ASD, which is known to be less developed in people with ASD. Psychological flexibility mediates the experience of psychological distress, for example depression, anxiety and stress, which are known to be highly prevalent in this population. Currently, there are mixed results in relation to effectiveness of CBT; very few researchers have measured the effectiveness of ACT to increase psychological flexibility in an adult ASD population and determine if this mediates a reduction in psychological distress.

PURPOSE OF THE STUDY This research will add to the knowledge about how ACT guided self-help can be adapted for adults with ASD. It will give results on how effective ACT guided self-help is in supporting adults with ASD, to increase psychological flexibility and reduce psychological distress. If guided ACT self-help intervention is effective; this will help increase access and availability of psychological intervention for people with ASD, specifically in relation to associated difficulties in social communication and interaction.

PRIMARY OBJECTIVE To examine whether an ACT bibliotherapy intervention, for adults with a diagnosis of ASD who experience psychological distress, increases psychological flexibility.

SECONDARY OBJECTIVE(S) To examine whether psychological flexibility mediates changes in; personally-identified therapeutic goals, increasing psychological wellbeing and decreasing anxiety, stress and depression.

STUDY DESIGN This is a repeated measures design, using a single case experimental design (SCED). Each participant with be asked to complete weekly measures and shortened measure every three days, please see the outcome measures section for more details of the measures and timeframes. Weekly data collection will last for approximately 10 weeks (baseline and intervention phase), with a two week and four week follow-up.

DATA ANALYSIS SCED data will be predominantly analysed using visual analysis. Data will be plotted onto graphs to analyse the direction of the data (trend), the "magnitude" (level) and the variability of the data (stability). To find out if change from pre and post scores is reliable, a Reliable Change Index (RCI) will be conducted. To determine if any change is clinically significant, a Clinically Significant Criterion (CSC) will be conducted. The data will be analysed at the University of Lincoln and Students home (via secured sites). The data will be analysed using Excel software. No interim analysis is planned for safety, efficacy or management purposes.

ELIGIBILITY:
Inclusion Criteria:

1. 18+ years old with a formal diagnosis of Autistic Spectrum Disorder, without a diagnosis if an Intellectual Disability.
2. To be over the age of 18 years.
3. Accessing Nottingham City Autism Service
4. Experiencing elevated anxiety, and / or stress, and /or depression and meet the clinical threshold or moderate on the Depression, Anxiety and Stress Scale.
5. Access to the internet via an electronic device (to complete electronic measures).
6. Agreement and knowledge of the time commitment for the completion of the intervention, competition of measure and change questionnaire at the end of the study.

Exclusion Criteria:

1. Unable to communicate fluently in English (justification: the cost of hiring an interpreter).
2. Unable to read English (justification: participant will be unable to read and engage in the bibliotherapy)
3. Adults who are currently accessing psychological therapy. If participants start psychological therapy during the study, they will be removed from the study (justification: unable to separate out effects of research intervention from psychological therapy intervention).
4. If they have a co-morbid diagnosis of intellectual disability (justification: may have different needs regarding therapy adaptations.
5. No access to mobile or internet (justification: unable to complete measures).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-01-20 (Estimated); Study Completion 2022-08-20 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Assessment of Acceptance and Commitment Therapy Process (CompACT) repeated measure of change | Administered pre-intervention phase, two week and four week post intervention
  23 Item measure of Psychological Flexibility
  The CompACT total score (out of 138). Higher scores indicate greater psychological flexibility (openness, awareness and activation)
  Th CompACT can also be separated into three subscales:
  1. Openness to Experince (OE) subscale (out of 60): Higher scores indicate greater openness to experience - i.e., willingness to experience internal events (thoughts, feelings, sensations, etc.) without trying to control or avoid them
  2. Behavioural Activation (BA) subscale (out of 30): Higher scores indicate greater behavioural awareness (mindful attention to current actions)
  3. Valued Action (VA) subscale (out of 48): Higher scores indicate greater engagement in valued actions (meaningful activity).
Comprehensive Assessment of Acceptance and Commitment Therapy Process (CompACT short form) repeated measure of change | Administered every three days during baseline and intervention period
  8 Item measure of Psychological Flexibility. Scores are derived by summing responses for each of the three subscales (Openness to Experience; Behavioural Awareness; Valued Action) or the scale as a whole (CompACT Total score).
  The full-scale CompACT Total score ranges from 0-48, with higher scores indicating greater psychological flexibility: The ability to attend and adapt to situational demands in the pursuit of personally meaningful longer-term goals.
  1. Openness to Experience (OE) subscale (0-18) higher scores indicating greater openness to experience (willingness to experience internal events [thoughts, feelings, sensations, etc.] without trying to control or avoid them).
  2. Behavioural Awareness (BA) subscale (0-12) higher scores indicating greater behavioural awareness (mindful attention to current actions).
  3. Valued Action (VA) subscale (0-18) with higher scores indicating greater engagement in valued actions (meaningful activity).
The Depression, Anxiety and Stress Scale (DASS-21) repeated measure of change | Administered as a screening questionaire; weekly during baseline and intervention phase, two and four weeks post intervention phase.
  21 Item measure of depression, stress and anxiety
  Scores for Depression, Anxiety and Stress are calculated by summing the scores for the relevant items. Recommended cut-off scores for conventional severity labels (normal, moderate, severe) are as follows:
  Depression: Normal 0-9, Mild 0-13, Moderate 14-20, Severe 21-27, Extremely Severe 28+
  Anxiety: Normal 0-7, Mild 8-9, Moderate -14, Severe 15-19, Extremely Severe 20+
  Stress: Normal 0-14, Mild 15-18, Moderate 19-25,Severe 26-33, Extremely Severe 37+

SECONDARY OUTCOMES:
Personal Questionnaire (PQ) repeated measure of change | Administered once during pre-intervention phase, Two and four weeks post intervention phase
  3 Item statements created by the client and based upon the clients values
  The Personal Questionnaire (PQ) is an expanded target complaint measure which is individualized for each client. It intended to be a list of problems or behaviours that the client wishes to work on during the intervention, stated in the client's own words.
  Clients rate each question on a likert scale scale (0-5), higher scores indicating more success/achievement at the target behaviour.
World Health Organisation Quality of Life Questionnaire (WHO-QoL- BRIEF) repeated measure of change | Administered pre-intervention, weekly during baseline and intervention phase, two and four week post intervention
  26 Item measure assessing Quality of Life.
  The WHOQOL-BREF produces a quality of life profile. It is possible to derive four domain scores; physical health (out of 35), psychological (out of 30), social relationships (out of 15) and environment (out of 40).
  There are also two items that are examined separately: question 1 asks about an individuals overall perception of quality of life and question 2 asks about an individuals overall perception of their health.
  The four domain scores denote an individuals perception of quality of life in each particular domain.
  Domain scores are scaled in a positive direction (i.e. higher scores denote higher quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: David Dawson, Principal Investigator — The University of Lincoln
Locations (1):
- Nottingham City Autisum Service, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
1. No individual participant data will be shared with researchers not named in this study.
  2. The results of the World Health Organisations Quality of Life Questionnaire (WHOQoL) will be shared anomalously with the World Health Organisation as stipulated by the organisation and specified in the participant consent form.
  3. Data collected will be collated and results will be written for publication. All participants will remain autonomous. The target journal identified is The Journal of Contextual and Behavioural Science.

REFERENCES:
- [Background] A-Tjak JG, Davis ML, Morina N, Powers MB, Smits JA, Emmelkamp PM. A meta-analysis of the efficacy of acceptance and commitment therapy for clinically relevant mental and physical health problems. Psychother Psychosom. 2015;84(1):30-6. doi: 10.1159/000365764. Epub 2014 Dec 24. PMID 25547522
- [Background] Hayes SC, Luoma JB, Bond FW, Masuda A, Lillis J. Acceptance and commitment therapy: model, processes and outcomes. Behav Res Ther. 2006 Jan;44(1):1-25. doi: 10.1016/j.brat.2005.06.006. PMID 16300724
- [Background] Hirvikoski T, Blomqvist M. High self-perceived stress and poor coping in intellectually able adults with autism spectrum disorder. Autism. 2015 Aug;19(6):752-7. doi: 10.1177/1362361314543530. Epub 2014 Jul 29. PMID 25073750
- [Background] Lane JD, Gast DL. Visual analysis in single case experimental design studies: brief review and guidelines. Neuropsychol Rehabil. 2014;24(3-4):445-63. doi: 10.1080/09602011.2013.815636. Epub 2013 Jul 24. PMID 23883189
- [Background] Lecavalier L. Behavioral and emotional problems in young people with pervasive developmental disorders: relative prevalence, effects of subject characteristics, and empirical classification. J Autism Dev Disord. 2006 Nov;36(8):1101-14. doi: 10.1007/s10803-006-0147-5. PMID 16897387
- [Background] Swain J, Hancock K, Hainsworth C, Bowman J. Acceptance and commitment therapy in the treatment of anxiety: a systematic review. Clin Psychol Rev. 2013 Dec;33(8):965-78. doi: 10.1016/j.cpr.2013.07.002. Epub 2013 Jul 16. PMID 23999201
- [Background] Weston L, Hodgekins J, Langdon PE. Effectiveness of cognitive behavioural therapy with people who have autistic spectrum disorders: A systematic review and meta-analysis. Clin Psychol Rev. 2016 Nov;49:41-54. doi: 10.1016/j.cpr.2016.08.001. Epub 2016 Aug 4. PMID 27592496
- [Background] Bruggink A., Huisman S., Vuijk R, Kraaij V, & Garnefski N. Cognitive emotion regulation, anxiety and depression in adults with autism spectrum disorder. Research in Autism Spectrum Disorders 22, 34-44, 2016
- [Background] Jacobson NS, Follette WC, & Revenstorf D. Psychotherapy outcome research: Methods for reporting variability and evaluating clinical significance. Behavior therapy 15(4):336-352, 1984.
- [Background] Cath DC, Ran N, Smit JH, van Balkom AJ, Comijs HC. Symptom overlap between autism spectrum disorder, generalized social anxiety disorder and obsessive-compulsive disorder in adults: a preliminary case-controlled study. Psychopathology. 2008;41(2):101-10. doi: 10.1159/000111555. Epub 2007 Nov 23. PMID 18033980

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-16): https://cdn.clinicaltrials.gov/large-docs/51/NCT04376151/Prot_SAP_000.pdf